CLINICAL TRIAL: NCT04542915
Title: COVID-19-Related Health and Practices Among Dental Hygienists
Status: Completed | Type: Observational
Sponsor: American Dental Association (Other)
Collaborators: American Dental Hygienists Association (Unknown)
Responsible Party: Principal Investigator, Cameron Estrich, Health research analyst, American Dental Association
Other Study IDs: ADA20-11
Record Dates: First submitted 2020-09-08; First posted 2020-09-09 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: SARS-CoV Infection; Anxiety; Depression; Occupational Problems; Severe Acute Respiratory Syndrome; Coronavirus Infection
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; Anxiety Disorders; Depression; Coronavirus Infections

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- U.S. licensed dental hygienists: Dental hygienists licensed in the United States. No intervention will be administered.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention.

SUMMARY:
As dental practices reopen their practices during a global pandemic, the risk of 2019 novel coronavirus (COVID-19) infection that dental hygienists face in providing dental care remains unknown. Estimating the occupational risk of COVID-19, and producing evidence on the types of infection control practices and dental practices that may affect COVID-19 risk, is therefore imperative. These findings could be used to describe the prevalence and incidence of COVID-19 among dental hygienists, determine what infection control steps dental hygienists take over time, describe dental hygienists' employment during the COVID-19 pandemic, and estimate whether infection control adherence in dental practice is related to COVID-19 incidence.

ELIGIBILITY:
Inclusion Criteria:

* Dental hygienist
* Licensed in the United States
* 18 years of age or older

Exclusion Criteria:

* Not employed as a dental hygienist as of March 1, 2020

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Dental hygienists licensed in the United States
Sampling Method: Non-Probability Sample
Enrollment: 6976 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
COVID-19 probable or confirmed case | 18 months
  2019 novel coronavirus (COVID-19) case as confirmed by clinician and/or detection of SARS-CoV-2 antigen or antibody

SECONDARY OUTCOMES:
Anxiety | 12 months
  Assessed using the Patient Health Questionnaire for Depression and Anxiety (PHQ-4). Two items scored 0 to 3 (total score of 0-6), with higher numbers indicating greater anxiety.
Depression | 12 months
  Assessed using the Patient Health Questionnaire for Depression and Anxiety (PHQ-4). Two items scored 0 to 3 (total score of 0-6), with higher numbers indicating greater depressive symptoms.
Dental practice infection control efforts | 12 months
  Self-reports of infection control efforts in the respondents' primary dental practices.
Personal protective equipment | 12 months
  Availability, frequency of use, and frequency of reuse of personal protective equipment
Employment status | 12 months
  Self-descriptions of current level of employment as a dental hygienist and reasons for non-employment.

CONTACTS AND LOCATIONS:
Locations (1):
- American Dental Association, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eldridge LA, Estrich CG, Gurenlian JR, Battrell A, Lynch A, Vujicic M, Morrissey R, Dershewitz S, Geisinger ML, Araujo MWB. US dental health care workers' mental health during the COVID-19 pandemic. J Am Dent Assoc. 2022 Aug;153(8):740-749. doi: 10.1016/j.adaj.2022.02.011. PMID 35902154
- [Derived] Estrich CG, Gurenlian JR, Battrell A, Bessner SK, Lynch A, Mikkelsen M, Morrissey R, Araujo MWB, Vujicic M. COVID-19 Prevalence and Related Practices among Dental Hygienists in the United States. J Dent Hyg. 2021 Feb;95(1):6-16. PMID 33627448